CLINICAL TRIAL: NCT01380314
Title: Treatment of Bolivian Cutaneous Leishmaniasis With a Combination of Oral Miltefosine Plus Topical Imiquimod 5%
Brief Title: Oral Miltefosine Plus Topical Imiquimod to Treat Cutaneous Leishmaniasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Foundation Fader (Other)
Responsible Party: Jaime Soto, Fundación Fader
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Bol-2008/01
Record Dates: First submitted 2008-05-07; First posted 2011-06-27 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Cutaneous Leishmaniasis
Keywords: leishmaniasis; cutaneois leishmaniasis; miltefosine; oral therapy; treatment; imiquimod
MeSH Terms: conditions — Leishmaniasis, Cutaneous; Leishmaniasis | interventions — miltefosine; Imiquimod

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Miltefosine 150 mg x day + Imiquimod 5%
  Interventions: Drug: Miltefosine + Imiquimod
- 2 (Placebo Comparator): Miltefosine 150 mg x day + Placebo
  Interventions: Drug: Miltefosine 150 mg x day + Placebo

INTERVENTIONS:
Drug: Miltefosine + Imiquimod — 150 mg x d during 28 days and cream applied every other day during 3 weeks
  Arms: 1
Drug: Miltefosine 150 mg x day + Placebo — 150 mg x d during 28 days and cream applied every other day during 3 weeks
  Arms: 2

SUMMARY:
Cutaneous leishmaniasis is endemic in the New World from approximately the US-Mexican border through Central America and the Northern part of South America down to the level of Rio de Janeiro.

Until recently, the standard treatment for the leishmaniases was pentavalent antimony (Glucantime or Pentostam). The cure rate for L panamensis in Colombia is 91%-93% [Soto, 1993; Velez, 1997], a large study with several formulations of antimony found a combined Bolivia-Colombia cure rate of 86% [Soto, 2004b], and in work just completed, the cure rate in Palos Blancos, Bolivia is 15 of 16 = 94% [ Soto, manuscript in preparation]. Nevertheless, pentavalent antimonials have the disadvantages of multiple injections and mild-moderate clinical toxicity [gastrointestinal complaints, liver enzyme elevations, pancreatic enzyme elevations], all of which are particularly unpleasant for a moderate clinical problem such as cutaneous leishmaniasis.

The oral agent Miltefosine has now been shown to be as effective as antimony in Colombia and Bolivia. In Colombia, the cure rate for miltefosine was 91% [Soto 2004a] and in the just-completed trial in Palos Blancos, the cure rate for miltefosine was 32 of 37 = 88 % . Side effects seen in patients with cutaneous disease that can be specifically attributed to the drug are nausea and vomiting of mild grade in approximately 25% of patients, and low-grade elevation of creatinine also in approximately 25% of patients [Soto 2001; Soto 2004].

The 6-month cure rate did not reach 100%, and miltefosine was relatively slow to cure compared to Sb. 31 of 44 evaluable miltefosine patients (70%) were cured by 1 month after therapy, compared to 16 of 16 evaluable Glucantime patients (100%).

Imiquimod (Aldara; 3M Pharmaceuticals) is a novel immune response-activating compound, approved by the FDA for cervical warts, that activates macrophage killing of Leishmania species. Combined imiquimod plus Glucantime was used as rescue treatment in 12 patients with Peruvian cutaneous leishmaniasis who had previously not responded to Glucantime alone. 90% of patients were cured at the 6-month follow-up period [Arevalo, 2001]. In a follow up study [Miranda-Verastegui et al, 2005], naïve patients were randomized between the combination of Sb plus imiquimod (18 patients) vs Sb plus placebo (20 patients). The cure rate at 1 month after therapy was 50% in the imiquimod +Sb group compared to 15% in the placebo+Sb group (p = 0.02). By 12 months after therapy, the Sb+placebo group had caught up, and the cure rate was 72%-75% in each group. Local side effects were evaluated. Edema, itching, burning, pain were equal in the two groups. There was more erythema in the imiquimod grup (55% of patients) compared to the placebo group (25% of patients).

The Imiquimod studies in neighboring Peru suggest that combination with this immunomodulator is capable of decreasing the time to cure, and potentially increasing the cure rate, in Andean cutaneous leishmaniasis. The present study will evaluate the combination of oral miltefosine plus topical imiquimod for cutaneous leishmaniasis in Bolivia. If in the first group of patients, cure rate at 1 month after therapy is appreciably above the 70% historic value for miltefosine alone and the cure rate at 6 months is greater than the 88% historic value for miltefosine alone, subsequent patients will be randomized between miltefosine+imiquimod and miltefosine+placebo cream.

ELIGIBILITY:
Inclusion Criteria:

* Gender: Male or female
* Age: >12 yrs of age
* Presentation: At least 1 lesion must be ulcerative. No more than 3 lesions. Parasitology: Parasitological confirmation of 1 lesion will be made by visualization or culture of leishmania from the biopsy or aspirate of the lesion.
* No specific or putatively specific therapy (Sb, pentamidine, amphotericin B, imidazoles, allopurinol) in the last 6 months

Exclusion Criteria:

* Previous treatment for leishmaniasis
* concomitant diseases by history
* abnormal complete blood counts (white blood count, hemoglobin, platelet count), values of liver transaminases (SGOT), kidney function tests (creatinine).
* pregnancy or breastfeeding or not willing to take contraception for 3 months after the end of treatment.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2008-03; Primary Completion 2010-03 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Healing of ulcers | 45 days

SECONDARY OUTCOMES:
Clinical findings and normal laboratory parameters | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Cenetrop, Santa Cruz, SC, Bolivia